CLINICAL TRIAL: NCT06324032
Title: EUS-Elastography and Contrast-Enhanced EUS Diagnostic Accuracy in the Differential Diagnosis of Subepithelial Gastrointestinal Tumors: a Multicenter Prospective Observational Study
Brief Title: SUNNYDAY: SUbepithelialgastroiNtestiNal Tumors Detection,accuracYDiAgnosis,ElastographY and Contrast-enhanced EUS
Acronym: SunnyDay021
Status: Recruiting | Type: Observational
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: 021-FPO20
Record Dates: First submitted 2024-02-15; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-02

CONDITIONS: Subepithelial Gastrointestinal Tumors
Keywords: subepithelial gastrointestinal tumors; Endoscopic Ultrasound; EUS; SETs; EUS Elastography; surgical resection; histopatological specimens
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with subepithelial gastrointestinal tumors: Patients with subepithelial gastrointestinal tumors
  Interventions: Procedure: EUS Elastography (EUS-E)

INTERVENTIONS:
Procedure: EUS Elastography (EUS-E) — All procedures will be performed with Olympus echoendoscopes (Olympus Europa SE & CO. KG, Hamburg, Germany) or Pentax echoendoscopes in combination with dedicated elastography software
  Other Names: Endoscopic Ultrasound (EUS); Contrast Enhanced-EUS (CE-EUS)

SUMMARY:
This will be a longitudinal, prospective, observational multicenter study where the role of EUS-E will be examined in differentiating subepithelial gastrointestinal tumors in 138 patients

DETAILED DESCRIPTION:
This will be a longitudinal, prospective, observational multicenter study that will enroll consecutive patients, with gastrointestinal SETs diagnosed by experienced endoscopists at Italian hospitals. This study will be conducted following the Helsinki Declaration after the approval by the ethics review board of all centers and will be recorded on Clinical-Trials.gov. All patients will provide their written informed consent for participating in the study. The EUS-E and CEUS analysis with SonoVue® will be performed during the same procedures. A subsequent diagnostic hypothesis on the nature of SETs will be formulated based on the B-mode, EUS-E, and CE-EUS characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with GI SETs scheduled for EUS-FNB 2 Patients with age > 18 but <85

Exclusion Criteria:

1. Patients with GI SETs <15mm
2. severe coagulopathy defined as abnormal prothrombin time (PT) or partial thromboplastin time (PTT) that does not normalize after administration of fresh frozen plasma
3. severe cardiopulmonary diseases and severe chronic kidney disease defined as
4. known allergic disposition to SonoVue®
5. pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: for patients with all types of Gastro Intestinal SETs.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of EUS-E accuracy qualitative | 4 weeks
  Evaluation of Endoscopic Ultrasound -Elastography (EUS-E)) accuracy (qualitative elastography) and contrast enhanced endoscopic ultrasound (CE-EUS) in the diagnosis of SETs compared to the histological data provided by the ultrasound-guided biopsy.
  the elastographic qualitative pattern will be assessed and described using an elastographic score.
  ELASTOGRAPHIC SCORE: three elastographic patterns will be used to define the stiffness of the SETs:
  * homogeneously green-pattern (soft)
  * mixed-type pattern (mild stiffness)
  * blue-predominant elastographic pattern (hard) Strain Ratio (SR) will be calculated by dividing the ROI placed on the normal GI wall at the periphery of the mass (ROI B) by the ROI placed on the lesion itself (ROI A). ROI A will be manually adjusted to cover the tumoral area as much as possible.
Evaluation of EUS-E accuracy quantitative | 4 weeks
  Evaluation of Endoscopic Ultrasound -Elastography (EUS-E) accuracy (quantitative elastography) and contrast enhanced endoscopic ultrasound (CE-EUS) in the diagnosis of SETs compared to the histological data provided by the ultrasound-guided biopsy.
  EUS-E compares the strain between the target area and other reference areas, to provide a semi-quantitative analysis of tissue stiffness.
  The SR (B/A quotients) will be calculated by the diagnostic US imaging system. The SRs will be measured and recorded 3 times in each procedure; the mean value will be considered as the final result for data analysis(to establish an SR cut-off to differentiate GIST from other SETs). Videos of 5 seconds will be recorded per each measurement.

SECONDARY OUTCOMES:
Evaluation of diagnostic accuracy of EUS-biopsy with fine needle biopsy (FNB) | 4 weeks
  Evaluation of diagnostic accuracy of Endoscopic Ultrasound biopsy (EUS-biopsy) with fine needle biopsy (FNB).
  Is obtained by evaluating the Strain Ratio (SR). Strain Ratio (SR) is a value resulting from the ratio between the stiffness of two user-defined areas within an elastogram ,which provides an objective evaluation of the hardness of lesion. Therefore, EUS-E has been applied to diseases of the pancreas, liver, prostate, lymphnodes, and other SETs
Evaluation of gene mutations in EUS-guided specimen | 24 weeks
  Evaluation of genetic mutations in ultrasound-guided endoscopic specimens by analyzing the tissue.
  All specimens will undergo histopathological examination, immunohistochemical evaluation, and molecular analysis
Correlation of elastographic and contrastographic characteristics of SETs with the pathological risk stratification. | 24 weeks
  Correlation of elastographic and contrastographic characteristics of SubEpithelial Tumors (SETs) with the pathological risk stratification.
  The elasticity of the tissues will be evaluated, which presents itself as a chromatic spectrum of shades and expressed graphically in an elastogram. The green color represents medium stiffness, blue reflects the hardest tissue and red the softest tissue.
Complication rate (perforations, bleeding) of the procedure | 48 hours
  Complication rate (perforations, bleeding) of the procedure will be obtained by evaluating the number of complications

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Staiano, MD, Principal Investigator — FPO-IRCCS di Candiolo
Locations (7):
- Italy (7):
  - Ospedale Santa Maria della Scaletta, Imola, Bologna
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Fondazione del Piemonte per l'Oncologia-IRCCS Candiolo, Candiolo, Turin,
  - Ospedale Humanitas Mater Domini, Castellanza, Varese
  - AOU Maggiore della Carità, Novara
  - Istituto Oncologico Veneto, Padua
  - AOU Città della Salute e della Scienza di Torino, Ospedale Molinette, Turin

IPD SHARING:
Plan to Share IPD: No
contact the principal investigator